CLINICAL TRIAL: NCT00432510
Title: Protocol LEVP2006-5: Pharmacokinetics of C1INH-nf in Hereditary Angioedema Subjects
Brief Title: Pharmacokinetics of C1 Esterase Inhibitor in Hereditary Angioedema Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LEVP2006-5
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; C1 esterase inhibitor (human)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Dose (Experimental): 1,000 Units (U) of C1INH-nf administered intravenously (IV).
  Interventions: Drug: C1 esterase inhibitor [human] (C1INH-nf)
- First Dose Followed by Second Dose (Experimental): 1,000 U of C1INH-nf administered IV, followed by a second 1,000 U dose 60 minutes later.
  Interventions: Drug: C1 esterase inhibitor [human] (C1INH-nf)

INTERVENTIONS:
Drug: C1 esterase inhibitor [human] (C1INH-nf)

SUMMARY:
The study objective was to describe the pharmacokinetics (PK) of one or two doses of C1 esterase inhibitor (C1INH-nf) in hereditary angioedema (HAE) subjects who were not experiencing an HAE attack.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in LEVP2005-1 (current or in the past)

Exclusion Criteria:

* C1 inhibitor infusion within the last 7 days
* Signs of any HAE attack
* HAE attack within 7 days before actual infusion of C1INH-nf
* Change in the dosage of androgens in the last 14 days before the study
* Use of antifibrinolytics in the last 7 days before the study
* Change in oral conceptive medication in the last two months before the study
* History of clinically relevant antibody development to C1 inhibitor
* Use of oral anticoagulant medication in the last 14 days
* Use of heparin within the last two days prior to the study
* History of allergic reaction to C1 inhibitor or other blood products
* Current participation (or within the past 90 days) in any investigational drug study other than those sponsored by Lev Pharmaceuticals
* Pregnancy or lactation
* B-cell malignancy
* Any clinically significant medical condition, such as renal failure, that in the opinion of the investigator would interfere with the subject's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-10-09 (Actual); Primary Completion 2007-02-28 (Actual); Study Completion 2007-02-28 (Actual)

PRIMARY OUTCOMES:
PK will be analyzed by means of incremental recovery, in vivo half-life, area under the curve, clearance, and mean residence time. | 1 week
C1 inhibitor (functional and antigenic) and C4 antigen serum levels will be measured at a United States Clinical Laboratory Improvement Amendments-certified laboratory and the research division of Sanquin Blood Supply Foundation. | 1 week

SECONDARY OUTCOMES:
Number and severity of adverse events. | 3 months
Change in clinical laboratory safety parameters from pre- to post-infusion. | 3 months
Change in vital signs from pre- to post-infusion. | 30 minutes (Single Dose), 90 minutes (First Dose Followed by Second Dose)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- United States (6):
  - University of California, San Diego, San Diego, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - Family Allergy and Asthma Center, Atlanta, Georgia
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Penn State University, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas